CLINICAL TRIAL: NCT04327765
Title: A Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetic Profile of Staccato Granisetron (AZ-010) in Healthy Volunteers
Brief Title: Staccato® Granisetron Multiple Dose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AMDC-010-102
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Cohort 1 (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: 0.5mg AZ-010
- Cohort 2 (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: 1mg AZ-010
- Cohort 3 (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: 3mg AZ-010

INTERVENTIONS:
Combination Product: 0.5mg AZ-010 — Subject will receive a single inhaled dose (0.5mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Placebo
  Arms: Cohort 1
Combination Product: 1mg AZ-010 — Subject will receive a single inhaled dose (1mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Placebo
  Arms: Cohort 2
Combination Product: 3mg AZ-010 — Subject will receive a single inhaled dose (3mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Placebo
  Arms: Cohort 3

SUMMARY:
To examine the tolerability and safety of AZ-010 following 7 days of dosing (up to 3 mg) in healthy volunteers To characterize the pharmacokinetics of AZ-010 following 7 days of dosing (up to 3 mg) in healthy volunteers

DETAILED DESCRIPTION:
A Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetic Profile of Staccato Granisetron (AZ-010) in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on a medical evaluation including history, physical examination, vital signs, electrocardiograms (ECGs) and laboratory tests assessed at the screening visit and prior to the first dose of study drug.
* Body weight ≥ 50 kg and BMI within the range of 18 to 32 kg/m2, inclusive, at screening.
* Negative urine tests for selected drugs of abuse and alcohol breath test at screening and Day 1.

Exclusion Criteria:

* Any significant medical condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 8 days
  Number of Subjects with Adverse Events as a measure of Safety and Tolerability

SECONDARY OUTCOMES:
Measurement of Granisetron Exposure in Plasma | 8 days
  AUC
Measurement of Granisetron Maximum exposure in Plasma | 8 days
  Cmax
Measurement of Granisetron Time to Maximum Exposure in Plasma | 8 days
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Terry O'Reilly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States